CLINICAL TRIAL: NCT00827398
Title: Treatment of Steroid Resistant Grade II to IV GVHD by Infusion MSCof Mesenchymal Stem Cells Expanded With Human Plasma and Platelet Lysate a Phase I/II Study
Brief Title: Treatment of Steroid Resistant GVHD by Infusion MSC
Acronym: MSCforGVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: N.M. Wulffraat (Other)
Responsible Party: Sponsor-Investigator, N.M. Wulffraat, MD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL13729.000.07
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2014-11-06 (Estimated); Status verified 2014-11

CONDITIONS: Graft-versus-host-disease
Keywords: MSC; GVHD; Adults; Children; steroid refractory acute GVHD occurring after allogeneic stem cell transplantation
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: MSC (hPPL) — Treatment with MSCs (hPPL) is indicated as soon as steroid refractory acute GVHD is diagnosed
  Other Names: Mesenchymal Stem Cells

SUMMARY:
For numerous malignant diseases allogeneic hematopoietic stem cell transplantation (HSCT) is the only curative therapy. One of the major complications is the occurrence of acute graft-versus-host-disease (aGVHD). Thirty to eighty percent of patients after HSCT develop aGVHD despite the prophylactic application of different immunosuppressive drugs.

The response rates to the conventional first line treatment are only 15-35%4. In case of a steroid refractory aGVHD different therapeutic strategies have been evaluated, but with no satisfactory results so far. The mortality of patients suffering from steroid refractory aGVHD remains at 75-80%. Therefore, it remains important to search for new therapeutical strategies for the treatment of aGVHD.

DETAILED DESCRIPTION:
For numerous malignant and non-malignant hematological diseases allogeneic hemato¬poietic stem cell transplantation (HSCT) is the only curative therapy. One of the major complications is the occurrence of acute graft-versus-host-disease (aGVHD). Thirty to eighty percent of patients after HSCT develop aGVHD despite the prophylactic application of different immunosuppressive drugs depending on risk factors such as HLA-match, donor relation, age etc.1-3.

First line therapy of aGVHD > grade I consists of steroids at a dose of 2 mg/kg. The response rates to this treatment are only 15-35%4. In case of a steroid refractory aGVHD different therapeutic strategies have been evaluated, but with no satisfactory results so far. The mortality of patients suffering from steroid refractory aGVHD remains at 75-80%, although numerous studies with different treatment strategies have been conducted2-5. Therefore, it remains important to search for new therapeutical strategies for the treatment of aGVHD.

The first patient to receive mismatched Mesenchymal Stem Cells was a twenty-year-old woman with acute myeloid leukemia treated with peripheral blood stem cells combined with MSC from her haploidentical father. Lazarus et al. reported on 46 patients who received HSCs and culture-expanded MSCs from HLA-identical siblings. Moderate to severe acute GvHD was observed in 28% of the patients, and chronic GvHD was seen in 61%. The two-year progression-free survival was observed in 53% of the patients. MSC infusion caused no acute or long-term MSC-associated adverse events.

Traditionally, for MSC isolation and expansion, fetal calf serum (FCS) supplemented media are used. The use of FCS has however several drawbacks and potential problems. We have therefore established a MSC culture protocol in animal serum free conditions using human platelet lysate and human plasma instead.

The present phase I/II study is designed to gather further insight into the clinical benefit in 50 patients (adults and children) with GvHD exerted by MSC expanded with human platelet lysate and plasma

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed acute grade II-IV GVHD or chronic GVHD with an acute pattern matching grade II-IV after allogeneic stem cell transplantation
* Patients must have received 2 mg/kg/day of prednisolon for at least 3 consecutive days and experience progression of GVHD or no response to at least 7 days of steroid treatment.
* In addition to steroids the patient has received either cyclosporin
* Written informed consent
* MSC donor must be HIV, HTLV, hepatitis BS antigen, HCV and HBC, Treponema Pallidum antibody negative. MSC donors can be mismatched related donor, third party matched or mismatched donor.

Exclusion Criteria:

* Patients with poor performance, not expected to survive 3 weeks.
* Donor Chimerism below 90%
* Active uncontrolled CMV, EBV or fungal infection

Ages: 1 Month to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
number of adverse events after infusion of MSC (hPPL) | 6 months
Number of severe infections after MSC infusion | 6 months

SECONDARY OUTCOMES:
Response of acute GVHD | 6 months
Determination of incidence of chronic GVHD | 6 months
Survival | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nico M Wulffraat, Principal Investigator — UMC Utrecht; Jurgen H Kuball, MD, Principal Investigator — UMC Utrecht
Locations (2):
- Netherlands (2):
  - UMC Utrecht, department of pediatrics, Utrecht
  - UMCU department of Haematology, Utrecht